CLINICAL TRIAL: NCT07060625
Title: The Effect of Semi-recumbent Position on Hypoxemia During the Recovery Period of General Anesthesia After Lung Segment/Lobe Surgery: a Single Center, Prospective, Real-world Study
Brief Title: The Effect of Semi-recumbent Position on Hypoxemia After Lung Segment/Lobe Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Hao Yang, post-doctoral, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: L24-629
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer (Diagnosis); Hypoxemia
MeSH Terms: conditions — Lung Neoplasms; Disease; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 308 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: Semi-recumbent position during anesthesia recovery
  Interventions: Behavioral: Semi-reclining position
- Non exposed group: Supine position during anesthesia recovery

INTERVENTIONS:
Behavioral: Semi-reclining position — During anesthesia recovery, the patient's position should be in a semi-recumbent position
  Groups: Exposure group

SUMMARY:
Thoracoscopic surgery is the most common surgical approach in thoracic surgery, which reduces surgical trauma and postoperative pain compared with open thoracotomy, but postoperative complications should not be overlooked, with hypoxemia being particularly prominent. Postoperative hypoxemia is highly prevalent among patients recovering from non-cardiac surgery, accounting for over one-third of all cases. Hypoxemia impairs wound healing and leads to other severe complications such as cerebral dysfunction, arrhythmia, and myocardial ischemia, all of which adversely affect postoperative recovery. Although oxygen therapy can prevent and treat hypoxemia, many patients still experience hypoxia in the post-anesthesia care unit (PACU). Numerous studies have investigated various ventilation techniques aimed at enhancing postoperative pulmonary function, but the benefits of protective ventilation strategies may be lost during emergence from anesthesia. Several other studies also indicate that intraoperative ventilation measures do not improve postoperative pulmonary function. The lack of evidence demonstrating the efficacy of oxygen therapy or protective ventilation techniques in treating postoperative hypoxemia underscores the need to explore alternative strategies. Patient positioning during emergence from anesthesia is associated with perioperative and postoperative complications. Although no consensus exists on the optimal patient position during emergence, the supine position is often favored by anesthesiologists due to its simplicity and ease of monitoring. However, the reduced functional residual capacity associated with the supine position tends to promote airway closure and diminish gas exchange.

DETAILED DESCRIPTION:
Thoracoscopic surgery is the most common surgical approach in thoracic surgery, which reduces surgical trauma and postoperative pain compared with open thoracotomy, but postoperative complications should not be overlooked, with hypoxemia being particularly prominent. Postoperative hypoxemia is highly prevalent among patients recovering from non-cardiac surgery, accounting for over one-third of all cases. Hypoxemia impairs wound healing and leads to other severe complications such as cerebral dysfunction, arrhythmia, and myocardial ischemia, all of which adversely affect postoperative recovery. Although oxygen therapy can prevent and treat hypoxemia, many patients still experience hypoxia in the post-anesthesia care unit (PACU). Numerous studies have investigated various ventilation techniques aimed at enhancing postoperative pulmonary function, but the benefits of protective ventilation strategies may be lost during emergence from anesthesia. Several other studies also indicate that intraoperative ventilation measures do not improve postoperative pulmonary function. The lack of evidence demonstrating the efficacy of oxygen therapy or protective ventilation techniques in treating postoperative hypoxemia underscores the need to explore alternative strategies. Patient positioning during emergence from anesthesia is associated with perioperative and postoperative complications. Although no consensus exists on the optimal patient position during emergence, the supine position is often favored by anesthesiologists due to its simplicity and ease of monitoring. However, the reduced functional residual capacity associated with the supine position tends to promote airway closure and diminish gas exchange. In contrast, the semi-recumbent position (SRP) has been shown to increase vital capacity by 10% to 15%, enhance functional lung volume and residual capacity, and improve diaphragmatic range of motion, thereby promoting lung expansion and gas exchange. Currently, only one study has found that in patients undergoing laparoscopic-assisted upper abdominal surgery, 30° SRP during anesthesia recovery can reduce the incidence of postoperative hypoxemia. Therefore, we conducted this real-world study to test the efficacy and optimal tilt angle of SRP in reducing hypoxemia during anesthesia recovery in a large sample of patients undergoing thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years old; Undergo thoracoscopic segment/lobectomy; American Society of Anesthesiologists (ASA) grade 1~3

Exclusion Criteria:

* Patients with mental or cognitive dysfunction who cannot communicate normally; Patients with tracheal catheters retained in ICU; Patients with cervical spondylosis, ankylosing spondylitis and other patients who cannot lift their upper body; Patients who have participated in other clinical trials; Patients who refuse to sign informed consent; Patients who have had chest surgery in the past.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thoracoscopic lobectomy and segmental resection
Sampling Method: Probability Sample
Enrollment: 308 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-PACU hypoxemia | Perioperative
  defined as SpO2 <90% for less than 60 seconds

SECONDARY OUTCOMES:
The incidence of severe hypoxemia | Perioperative
  SpO2<75% or SpO2<90% lasting for more than 60 seconds at any time
the time of the first episode of hypoxemia | Perioperative
Airway first aid | Perioperative
  Defined as the need for jaw support to open the airway, mask noninvasive positive pressure ventilation, or pharyngeal or nasopharyngeal airway assisted ventilation, reintubulation or laryngoscope placement
Breathing comfort | Perioperative
  Use a digital rating scale ranging from 0 to 10, with higher scores indicating greater comfort
Wound pain VAS score | measured and recorded at rest and cough, 5 and 30 minutes after extubation, before leaving PACU and 24,48 and 72 hours postoperative
blood gas analysis | Perioperative
The duration of PACU stay | Perioperative
Heart rate | Upon admission, before induction, after intubation, immediately after the end of surgery, immediately before extubation, immediately after admission to PACU and adjustment of position, 10 minutes after admission to PACU, and upon departure from PACU
Mean arterial pressure | Upon admission, before induction, after intubation, immediately after the end of surgery, immediately before extubation, immediately after admission to PACU and adjustment of position, 10 minutes after admission to PACU, and upon departure from PACU

OTHER OUTCOMES:
Adverse events related to position | Perioperative
  hypotension, arrhythmia
15-item recovery quality scale (Quality of Recovery-15, QoR-15) scores | at 1 and 3 days postoperative
Postoperative inflammatory markers | On the first day after surgery
  C-reactive protein, absolute value of neutrophils, absolute value of lymphocytes, absolute value of monocytes, white blood cell count, platelet count
length of hospital stay | 3-5 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yang Hao, postdoctor, Study Director
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No